CLINICAL TRIAL: NCT06075589
Title: Promoting Adjustment in Uveal Melanoma Survivorship: A Randomized Trial Targeting Illness Perceptions
Brief Title: Psychoeducation for Uveal Melanoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-000414
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Educational Status; Methods; Health Promotion; Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Participants watch two fifteen-minute educational videos and receive a mental health resource information sheet on study.
  Interventions: Behavioral: Education for Intervention
- Arm II (Experimental): Patients receive enhanced treatment as usual and receive a mental health resource information sheet on study.
  Interventions: Behavioral: Best Practice

INTERVENTIONS:
Behavioral: Education for Intervention — Participants watch two fifteen-minute educational videos and receive a mental health resource information sheet on study.
  Other Names: Health Promotion and Education; Questionnaire Administration
  Arms: Arm 1
Behavioral: Best Practice — Patients receive enhanced treatment as usual and receive a mental health resource information sheet on study.
  Arms: Arm II

SUMMARY:
This clinical trial evaluates a video-based psychoeducational intervention for patients with uveal melanoma. Uveal melanoma (UM) is a rare intraocular cancer. UM patients face an uncertain course of survivorship in terms of their visual acuity, treatment-related side effects, and risk for eventual metastasis of the cancer. Learning about patients' thoughts and reactions to informational resources may better support patients during ocular melanoma survivorship.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the efficacy of the psychoeducation intervention (compared to the control condition) in modifying illness perceptions of disease control, chronicity, and coherence (i.e., to become less threatening) over the course of the follow-up period.

SECONDARY OBJECTIVE:

I. To assess the efficacy of the psychoeducation intervention (compared to the control condition) in reducing the degree of participant's depressive and anxiety symptoms over the course of the follow-up period.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants watch two fifteen-minute educational videos and receive a mental health resource information sheet on study.

ARM II: Patients receive enhanced treatment as usual and receive a mental health resource information sheet on study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age 18 years and older at visit 1)
* History of uveal melanoma as documented in their University of California, Los Angeles (UCLA) medical record
* Receipt of uveal melanoma treatment and/or ongoing follow-up care at the UCLA Jules Stein Eye Institute, as documented in their UCLA medical record
* Ability to read, write, and converse in English
* Access to the internet via a computer or cell phone
* Access to a personal email address
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in illness perceptions of disease control | From baseline to day 77
  Will be assessed using the Brief Illness Perception Questionnaire (BIPQ) and will be examined across treatment and control conditions using multilevel models.
Change in illness perceptions of chronicity | From baseline to day 77
  Will be assessed using the BIPQ will be examined across treatment and control conditions using multilevel models.
Change in illness perceptions of coherence | From baseline to day 77
  Will be assessed using the BIPQ will be examined across treatment and control conditions using multilevel models.

SECONDARY OUTCOMES:
Domains of mental health: Anxiety | From baseline to day 77
  Will be assessed by multilevel models of anxiety symptoms as functions of treatment condition (i.e., group assignment). Anxiety symptoms will be assessed at all assessment points with the Generalized Anxiety Disorder Scale-7.
Domains of mental health: Depression | From baseline to day 77
  Will be assessed by multilevel models of depression symptoms as functions of treatment condition (i.e., group assignment). Depressive symptoms will be assessed at all assessment points with the well-validated 20-item Center for Epidemiologic Studies-Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anette Stanton, PhD, Principal Investigator — University of Califonia at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No